CLINICAL TRIAL: NCT06673680
Title: Role Of Colposcopy In Evaluation Of Suspicious Cervix
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omar Kamal Mohamed, Resident, Sohag University
Other Study IDs: colposcopy in cancer cervix
Record Dates: First submitted 2024-10-23; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cancer Cervix
Keywords: screening in cancer cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- colposcopic evaluation: do colposcopy and cervical punch biopsy then compare between findings
  Interventions: Device: Do colposcopy and cervical punch biopsy then compare between findings

INTERVENTIONS:
Device: Do colposcopy and cervical punch biopsy then compare between findings — The aim of this study is to correlate colposcopy and histopathological findings in early screening of suspicious cervix and cervical cancer. And to do a colposcopic evaluation of all cervical lesions and the early detection of all cervical precancer and invasive lesions of the cervix in symptomatic women.

SUMMARY:
do colposcopy and cervical punch biopsy then compare between findings

DETAILED DESCRIPTION:
The aim of this study is to correlate colposcopy and histopathological findings in early screening of suspicious cervix and cervical cancer. And to do a colposcopic evaluation of all cervical lesions and the early detection of all cervical precancer and invasive lesions of the cervix in symptomatic women.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 64 years old.
* Women with symptoms such as white discharge, post-coital bleeding, and intermenstrual bleeding.
* Women with the clinically unhealthy cervix (erosion, bleeding on touch, simple leukoplakia, keratinization)
* Women with Pap smear showing dysplasia

Exclusion Criteria:

* Pregnant women
* Women having active vaginal bleeding.
* Any past treatment for cervical lesions.
* Women having frank growth of cervix.
* Women who underwent a hysterectomy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — study use colposcope in screening of cancer cervix
Study Population: * Age from 30 to 64 years old.
  * Women with symptoms such as white discharge, post-coital bleeding, and intermenstrual bleeding.
  * Women with the clinically unhealthy cervix (erosion, bleeding on touch, simple leukoplakia, keratinization)
  * Women with Pap smear showing dysplasia.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
comparison between colposcopic findings of suspicious cervix and histopathologic findings | baseline
  Correlate colposcopy and histopathological findings in early screening of suspicious cervix and cervical cancer. And to do a colposcopic evaluation of all cervical lesions and the early detection of all cervical precancer and invasive lesions of the cervix in symptomatic women.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem A prof, MD, Study Director — Sohag university hospitals
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No